CLINICAL TRIAL: NCT00293423
Title: Phase I/II Trial of Heat Shock Protein Peptide Complex-96 (HSPPC-96) Vaccine for Patients With Recurrent High Grade Glioma
Brief Title: GP96 Heat Shock Protein-Peptide Complex Vaccine in Treating Patients With Recurrent or Progressive Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Agenus Inc. (Industry); American Brain Tumor Association (Other)
Responsible Party: Principal Investigator, Orin Bloch, MD, Principal Investigator, University of California, San Francisco
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 05103; UCSF-H41995-27311-01 (Other: University of California, San Francisco); NCI-2011-01231 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP)); P50CA097257-06 (NIH); R01CA164714-02 (NIH)
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Brain Neoplasms | interventions — vitespin; Heat-Shock Response; myelin oligodendrocyte glycoprotein (74-96), human; glucose-regulated proteins; Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Vaccine (Experimental): Patients received 25 micrograms of HSPPC-96 bi-weekly or weekly for the first 4 vaccinations followed by biweekly injections.
  Interventions: Biological: HSPPC-96; Procedure: Standard Surgical Resection
- Phase 2: Vaccine (Experimental): Treatment consisted of 25 mcg of HSPPC-96 weekly for at least 4 weeks, followed by biweekly injections (pending vaccine availability) for up to 52 weeks from the date of surgical resection.
  Interventions: Biological: HSPPC-96; Procedure: Standard Surgical Resection

INTERVENTIONS:
Biological: HSPPC-96 — 25 mcg
  Other Names: Heat Shock; Glycoprotein 96; Gp96
Procedure: Standard Surgical Resection — Patients will undergo standard surgical resection of intracranial tumor
  Other Names: Craniotomy

SUMMARY:
Vaccines made from a person's tumor cells, such as gp96 heat shock protein-peptide complex, may help the body build an effective immune response to kill tumor cells. This phase I/II trial is studying the side effects and best dose of gp96 heat shock protein-peptide complex vaccine to see how well it works in treating patients with recurrent or progressive high-grade glioma over time.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

* Phase 1: [closed to accrual as of 7/25/2007]: Determine the safety and best tolerated dose and frequency of gp96 heat shock protein-peptide complex vaccine in patients with recurrent or progressive high-grade glioma.
* Phase 2: Determine the clinical response to treatment, time to disease recurrence and progression, and overall survival of patients treated with this vaccine.

SECONDARY OBJECTIVES:

* Determine the immune response in patients treated with this vaccine.
* Determine survival outcomes in patients treated with this vaccine.

OUTLINE: This is a dose-escalation, phase I study (closed to accrual as of 7/25/2007) followed by a phase II study.

PHASE I [closed to accrual as of 7/25/2007]:

Patients underwent surgical resection. Viable tumor tissue is used to generate the gp96 heat shock protein-peptide complex (HSPPC-96) vaccine. Patients with primary disease receive standard adjuvant therapy after surgery. Patients whose disease progresses during or after standard adjuvant therapy receive the HSPPC-96 vaccine. Patients with recurrent disease receive the HSPPC-96 vaccine between 2-8 weeks after surgery. The HSPPC-96 vaccine is administered intradermally every 1-3 weeks for at least 4 doses and then every 2-3 weeks thereafter in the absence of disease progression, unacceptable toxicity, or vaccine depletion. Cohorts of 6 patients received the HSPPC-96 vaccine at escalating dose frequencies until the maximum tolerated dose (MTD) was determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experienced a dose-limiting toxicity.

PHASE II: Patients received the HSPPC-96 vaccine as in phase I at the appropriate dose frequency determined in phase I (closed to accrual as of 7/25/2007). The HSPPC-96 vaccine is administered intradermally every 1-3 weeks for at least 4 doses and then every 2 weeks thereafter in the absence of disease progression, unacceptable toxicity, or vaccine depletion. After completion of study treatment, patients are followed periodically until death, lost to follow-up, or end of study.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant recurrent glioma*, including any of the following:

  * Glioblastoma

    * Glioblastoma multiforme
* Recurrent disease or progressive primary disease
* Surgically accessible tumor for which surgical resection is indicated and has not been previously irradiated
* Prior radiotherapy required
* No prior oncophage therapy or immunotherapy for glioma

PATIENT CHARACTERISTICS:

* Karnofsky performance status 80-100%
* Life expectancy ≥ 8 weeks
* Absolute granulocyte count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Alkaline phosphatase and serum glutamic-pyruvic transaminase (SGPT) <=2.5 times normal
* Bilirubin < 1.5 mg/dL
* Blood Urea Nitrogen (BUN) < 1.5 times normal OR creatinine < 1.5 times normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for at least 4 weeks after completion of study treatment
* No uncontrolled active infection
* No bleeding diathesis
* No psychiatric or medical situation that would preclude study compliance
* No unstable or severe concurrent medical condition
* No other cancer or concurrent malignancy within the past 5 years except adequately treated nonmetastatic in situ carcinoma of the uterine cervix, nonmetastatic nonmelanoma skin cancer, or in complete remission and off all therapy for that disease
* No systemic autoimmune disease (e.g., Hashimoto's thyroiditis) and/or any history of primary or secondary immunodeficiency

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 2 weeks since prior vincristine
* At least 6 weeks since prior nitrosoureas
* At least 4 weeks since prior temozolomide or other cytotoxic chemotherapy
* At least 4 weeks since prior investigational agents
* At least 1 week since prior noncytotoxic agents
* At least 3 weeks since prior procarbazine
* No radiotherapy within the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-11-18 (Actual); Primary Completion 2013-01-12 (Actual); Study Completion 2013-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Clarke, MD, Study Chair — University of California, San Francisco
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Columbia University, New York, New York
  - University Hospitals Case Medical Center, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crane CA, Han SJ, Ahn B, Oehlke J, Kivett V, Fedoroff A, Butowski N, Chang SM, Clarke J, Berger MS, McDermott MW, Prados MD, Parsa AT. Individual patient-specific immunity against high-grade glioma after vaccination with autologous tumor derived peptides bound to the 96 KD chaperone protein. Clin Cancer Res. 2013 Jan 1;19(1):205-14. doi: 10.1158/1078-0432.CCR-11-3358. Epub 2012 Aug 7. PMID 22872572
- [Result] Bloch O, Crane CA, Fuks Y, Kaur R, Aghi MK, Berger MS, Butowski NA, Chang SM, Clarke JL, McDermott MW, Prados MD, Sloan AE, Bruce JN, Parsa AT. Heat-shock protein peptide complex-96 vaccination for recurrent glioblastoma: a phase II, single-arm trial. Neuro Oncol. 2014 Jan;16(2):274-9. doi: 10.1093/neuonc/not203. Epub 2013 Dec 12. PMID 24335700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase 1 Recruitment took place between August 11, 2005 and July 25, 2007 for participants scheduled for gross total resection of recurrent Glioblastoma multiforme (GBM)
  Phase 2 Recruitment took place between October 3, 2007 and October 24, 2011 for participants scheduled for gross total resection of recurrent Glioblastoma multiforme (GBM)
Period: Surgical Resection
Arm/Group | Phase 1: Vaccine | Phase 2: Vaccine
Started | 28 | 68
Completed (All patients underwent aggressive resection with intra-operative collection of tissue to generate autologous vaccine. Only participants with adequate tissue collected to generate enough vaccine and whose vaccines passed quality control standards received the vaccine and constituted the intent-to-treat group) | 12 | 41
Not Completed | 16 | 27
Not completed — Less than a 90% extent of resection | 0 | 1
Not completed — Postoperative Karnofsky Performance Score <70% | 0 | 4
Not completed — Insufficient tumor obtained to generate vaccine | 9 | 13
Not completed — disease progression prior to initial vaccination | 2 | 9
Not completed — processing error during surgical resection | 1 | 0
Not completed — Withdrawal by Subject | 4 | 0
Period: Vaccination Treatment Period
Arm/Group | Phase 1: Vaccine | Phase 2: Vaccine
Started | 12 | 41
Completed | 12 | 38
Not Completed | 0 | 3
Not completed — Received < 4 required vaccinations | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Vaccine | Phase 2: Vaccine | Total
Number analyzed (Participants) | 28 | 68 | 96
Age, Customized [Count of Participants; unit: Participants]
  20-29 years old | 0 | 3 | 3
  30-39 years old | 3 | 2 | 5
  40-49 years old | 5 | 14 | 19
  50-59 years old | 12 | 23 | 35
  60-69 years old | 6 | 20 | 26
  70-79 years old | 2 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 19 | 32
  Male | 15 | 49 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 28 | 68 | 96
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 27 | 65 | 92
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 28 | 68 | 96
Median Number of Vaccine Doses Administered [Median (Full Range); unit: vaccine injections] — Population: Vaccines were only given to the intent-to-treat population
  vaccine injections
    number analyzed (Participants) | 12 | 41 | 53
    (all) | 6 [4 to 22] | 6 [1 to 15] | 6 [1 to 22]

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) (Phase 1)
Description: MTD determination will be based on the occurrence of dose-limiting toxicities. The MTD will be 1 dose below the dose that defined the dose-limiting toxicities
Time Frame: Up to 4 weeks
Measure: Number; unit: micrograms
Arm/Group | Phase 1: Vaccine
Number analyzed (Participants) | 12
micrograms | 25

2. Primary Outcome: Frequency of gp96 Heat Shock Protein-peptide Complex Vaccine (Phase 1)
Description: The frequency of dosing of the first 4 injections to be recommended for Phase 2 will be determined by reviewing the reported number of dose-limiting toxicities for weekly or bi-weekly injections.
Time Frame: Up to 6 months
Measure: Number; unit: weeks between doses
Arm/Group | Phase 1: Vaccine
Number analyzed (Participants) | 12
weeks between doses | 2

3. Primary Outcome: Number of Participants With Dose Limiting Toxicities (Phase 1)
Description: Systemic toxicity will be graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.0. Dose-limiting toxicity is defined as any of the following that are attributable to vaccine therapy: Any grade 3, 4 or 5 toxicity, Any grade >=2 clinical autoimmunity with the potential to threaten critical organs (including lungs, heart, kidney, bowel, bone marrow, liver or central nervous system (CNS), or eyes), and any removal of a patient from therapy due to toxicity
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: Vaccine
Number analyzed (Participants) | 12
Participants | 0

4. Primary Outcome: Median Progression-free Survival at 6 Months (Phase 2)
Time Frame: 6 months
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Vaccine
Number analyzed (Participants) | 41
weeks | 19.1 [14.1 to 24.1]

5. Primary Outcome: Percentage of Participants With Progression-free Survival at 12 Months (Phase 2)
Description: Defined as the percentage of participants with confirmed response and who have not progressed from date of surgical resection until death or censored at 12 months
Time Frame: Up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Vaccine
Number analyzed (Participants) | 41
percentage of participants | 29.3 [16.6 to 45.7]

6. Secondary Outcome: Number of Patients With an Immunological Response (Phase 1)
Description: An immunological response is defined as an absolute lymphocyte count (ALC) less than the lower limit of normal (1.0 × 109cells/L), according to the standard laboratory reference range
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Phase 1: Vaccine
Number analyzed (Participants) | 12
participants | 11

7. Secondary Outcome: Number of Patients With an Immunological Response (Phase 2)
Description: as for outcome 6
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Vaccine
Number analyzed (Participants) | 41
Participants | 27

8. Secondary Outcome: Number of Participants With Grade 3 or Higher, Vaccine Treatment-Related Adverse Events by Toxicity (Phase 2)
Description: Vaccine treatment-related Adverse Events with a grade >=3 according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4 will be reported.
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Phase 2: Vaccine
Number analyzed (Participants) | 41
participants | 1

9. Secondary Outcome: Median Overall Survival (Phase 2)
Description: Overall survival is defined as the length of time from date of surgical resection until death or censored at end of study period
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Phase 2: Vaccine
Number analyzed (Participants) | 38
weeks | 42.6 [34.7 to 50.5]

10. Secondary Outcome: Percentage of Participants Surviving at 6 Months (Phase 2)
Description: Defined as the percentage of participants still alive from date of surgical resection until death or censored at 6 months
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Vaccine
Number analyzed (Participants) | 38
percentage of participants | 90.2 [75.9 to 96.8]

11. Secondary Outcome: Percentage of Participants Surviving at 12 Months (Phase 2)
Description: Defined as the percentage of participants still alive from date of surgical resection until death or censored at 12 months
Time Frame: Up to 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Vaccine
Number analyzed (Participants) | 38
percentage of participants | 29.3 [16.6 to 45.7]

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | Phase 1: Vaccine | Phase 2: Vaccine
All-Cause Mortality (participants affected / at risk) | 0/12 | 39/41
Serious Adverse Events (participants affected / at risk) | 0/12 | 8/41
Other Adverse Events (participants affected / at risk) | 12/12 | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Vaccine (N=12) | Phase 2: Vaccine (N=41)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Wound (Infections and infestations) | 0 | 1
Neurology - Other (Nervous system disorders) | 0 | 1
Psychiatric disorders - Other (Psychiatric disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Peripheral Motor Neuropathy (Nervous system disorders) | 0 | 1
Skin Infection (Cellulitis) (Infections and infestations) | 0 | 1
Infections and infestations - Other, Appendix (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Vaccine (N=12) | Phase 2: Vaccine (N=41)
Vascular (Vascular disorders) | 0 (0) | 3 (41)
Hematoma (Vascular disorders) | 0 (0) | 3 (3)
Cerebrospinal fluid leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (6)
Seizure (Nervous system disorders) | 4 (9) | 6 (6)
Mood (Psychiatric disorders) | 1 (1) | 7 (7)
Hydrocephalus (Nervous system disorders) | 0 (0) | 3 (3)
Focal deficit (Investigations) | 0 (0) | 28 (28)
Cognitive (General disorders) | 2 (2) | 20 (20)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 5 (8) | 9 (9)
Metabolic (Metabolism and nutrition disorders) | 9 (32) | 16 (16)
Lymphatic (Blood and lymphatic system disorders) | 2 (2) | 5 (5)
Infection (Infections and infestations) | 1 (1) | 11 (11)
Leukopenia (Blood and lymphatic system disorders) | 4 (9) | 10 (10)
Coagulopathy (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
Genitourinary/renal (Renal and urinary disorders) | 2 (2) | 8 (8)
Gastrointestinal (Gastrointestinal disorders) | 4 (12) | 14 (14)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5)
Injection site reaction (Investigations) | 6 (9) | 17 (17)
Fever (General disorders) | 0 (0) | 4 (4)
Fatigue (General disorders) | 7 (10) | 12 (12)
Anorexia (General disorders) | 1 (2) | 4 (4)
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ocular/Visual - Other (Eye disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes